CLINICAL TRIAL: NCT06400576
Title: Effects of Smartphone and Headphone Usage on Baropodometric Parameters in Healthy Individuals
Brief Title: Smartphone & Headphone Effects on Baropodometric Parameters
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Assist, Prof, Hacettepe University
Other Study IDs: SPP
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Smartphone Addiction; Postural; Defect; Dual Task
Keywords: Postural oscillation; Headphone use; Messaging; Balance; Gait; Foot Pressure Distrubition; Smartphone addiction; Daily activites
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Headphone and Smartphone Usage Group: The group where participants listen to music while messaging and also where these activities are evaluated separately. The only group in the study.
  Interventions: Other: Headphone and Smartphone Intervention

INTERVENTIONS:
Other: Headphone and Smartphone Intervention — Asessment of participants' static balance and pressure distrubiton, posturographic balance and dynamic balance whilst using headphones and messaging.
  Other Names: FreeMed Baropodometric Device

SUMMARY:
The goal of this observational study is to observe baropodometric parameters such as postural sway and foot pressure distrubiton in healthy young participants between the ages of 18-35. The main questions it aims to answer are:

* How does headphone usage affect baropodometric parameters in healthy young individuals?
* How does texting affect baropodometric parameters in healthy young individuals?
* How does headphone usage while texting affect baropodometric parameters in healthy young individuals?

Participants will:

* Only be evaluated once.
* Stand on the Baropodometric device platform while standing, texting, listening to music, texting while listening to music for the static and posturographic balance evaluation.
* Walk on the baropdometric device platform while standing, texting, listening to music, texting while listening to music for dynamic evaluation.

DETAILED DESCRIPTION:
During our daily lives, the individuals perform many functions simultaneously. Two devices that modern technology has brought us are headphones and mobile phones, both of which are commonly used. Studies have shown that posture oscillation changes during walking while using a phone, but same studies also stated that more comprehensive studies are needed. There is no study in the literature that examines postural oscillation and foot pressure distribution while listening to music with headphones and messaging. The aim of this observational study is to evaluate the postural oscillation and foot pressure distribution during headphone use and messaging in healthy participants aged 18-35. The sample size of 35 participants was determined based on a similar study example using G-Power analysis. Participants will be assesed at Hacettepe University, Faculty of Physical Therapy and Rehabilitation. Participants will be selected based on eligibility criteria, and there will be only one group in the study; therefore, randomization will not be performed. Participants enrolled in the study will be evaluated using the FreeMED force platform (Sensor Medica, Italy). The platform itself is 40x40 cm in size and comes with two plates, each one meter long. When all components are assembled, a continuous surface of 2.4 meters is obtained. Participants will participate in static, posturographic, and dynamic evaluations. In each evaluation, participants will first stand still, then put on headphones and listen to music at 80 decibels with a tempo of 130 bpm, then type a message, and finally type a message while listening to music. Static evaluation will provide information about foot pressure distribution; posturographic evaluation will include Romberg tests with eyes open, eyes closed, standing on one foot, and standing on two feet; and dynamic evaluation will assess participants' walking phases and speed. The statistical analysis of the study will be performed using SPSS 23.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study voluntarily,
* Being between the ages of 18-35

Exclusion Criteria:

* Not agreeing to participate in the study voluntarily.
* Having a congenital spinal cord anomaly
* Existing neurological, orthopedic, inflammatory, cardiovascular, rheumatological, vestibular problems
* Having a surgical history of the spinal region

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young people who are volunteering to participate the study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Baropodometer assessments- Static pressure distribution | through study intervention, an average of 15 minutes
  Pressure distribution will be assessed with FreeMed baropodometric platform and the recording measurement unit will be percentages.
Baropodometer assessments- Posturographic center of gravity | through study intervention, an average of 15 minutes
  Center of gravity will be assessed with FreeMed baropodometric platform and the recording measurement unit will be milimeters.
Baropodometer assessments- Posturographic oscillations | through study intervention, an average of 15 minutes
  Oscillations will be assessed with FreeMed baropodometric platform and the recording measurement unit will be milimeters.
Baropodometer assesments - Posturographic Sway Length | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and the recording measurement unit will be milimeters.
Baropodometer assesments - Posturographic Displacement Towards X and Y axis | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and the recording measurement unit will be milimeters.
Baropodometer assessments- Posturographic average sway velocity | through study intervention, an average of 15 minutes
  Sway velocity will be assessed with FreeMed baropodometric platform and the recording measurement unit will be degrees.
Baropodometer assessments- Dynamic average surface | through study intervention, an average of 15 minutes
  Average surface will be assessed with FreeMed baropodometric platform and the recording measurement unit will be cm.
Baropodometer assessments- Dynamic average speed | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and the recording measurement unit will be milimeters/second.
Baropodometer assesments - Dynamic Gait Phase Durations | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and the recording measurement unit will be percentages
Feet Loading Pattern - Dynamic Longitudinal Arc | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and will be used to asses the feet loading pattern.
Feet Loading Pattern - Forefoot Reatfoot Load | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and will be used to asses the feet loading pattern.
Feet Loading Pattern - Medial Lateral Load | through study intervention, an average of 15 minutes
  It will be assessed with FreeMed baropodometric platform and will be used to asses the feet loading pattern.

SECONDARY OUTCOMES:
Forward Head Posture | At Baseline
  It will be assessed with a digital inclinometer, the measurement unit will be in degrees.
New York Posture Assesment | At Baseline
  This form will assess participants' postural alignment. Total scores range from 13 to 65, with results categorized as: 'excellent' (above 45), 'good' (40-44), 'fair' (30-39), 'poor' (20-29), and 'very poor'.
International Physical Activity Questionnaire | At Baseline
  This form will assess participants' physical fitness and well-being. Based on MET minutes per week, the results are categorized into three activity levels: inactive, minimally active and very active.
The Cognitive Flexibility Inventory | At Baseline
  The Cognitive Flexibility Inventory is a 20-item self-report measure to monitor how often individuals engaged in cognitive behavioural thought challenging interventions. The total score ranges between 20 and 140, where higher scores indicate more cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Cetin, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hatice Cetin, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No